CLINICAL TRIAL: NCT00450073
Title: Desktop Tanning Unit to Improve Vitamin D Status in Patients With Cystic Fibrosis and Short Bowel Syndrome: A Pilot Study
Brief Title: Improving Vitamin D Status In Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Associate Professor, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cystic Fibrosis Vitamin D
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D3 (Active Comparator): Vitamin D3=cholecalciferol 50,000 IU weekly
  Interventions: Drug: Vitamin D3
- vitamin D2 (Active Comparator): The intervention is an oral tablet of vitamin D2 (ergocaliferol 50,000 IU weekly) for 12 weeks.
  Interventions: Drug: ergocalciferol (vitamin D2)
- Sunlamp (Active Comparator): The intervention is the use of a Sunlamp (Sperti) to the skin 5 times a week for 12 weeks
  Interventions: Device: Sperti Del Sol Lamp

INTERVENTIONS:
Drug: ergocalciferol (vitamin D2) — 50,000 IU weekly
  Other Names: D2
  Arms: vitamin D2
Device: Sperti Del Sol Lamp — 5 times a week for 12 weeks
  Arms: Sunlamp
Drug: Vitamin D3 — 50,000 IU weekly
  Other Names: D3
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is to establish an effective method to correct vitamin D deficiency in subjects with cystic fibrosis. The investigators will examine cholecalciferol, ergocalciferol and UV light.

DETAILED DESCRIPTION:
Hypothesis of this study: Our hypothesis is that other methods such as cholecalciferol replacement and/or low dose ultraviolet radiation to the skin may be more effective in raising serum 25-hydroxyvitamin D levels than conventional ergocalciferol therapy.

Experimental strategy: We will conduct a prospective randomized trail to determine which recommended vitamin D therapy (tanning device, cholecalciferol or ergocalciferol) is effective in maintaining or improving vitamin D status during the winter months. We will recruit CF patients according to the following inclusion and exclusion criteria:

Inclusion: Subjects seen initially at the Emory CF center between the months of September and December, age >16, both males and females, confirmed cystic fibrosis by genetic testing or sweat testing, FEV1 >40%.

Exclusion: History of lung transplant or awaiting lung transplantation, current hospitalization or greater than 6 hospitalizations/year, history of malignancy, renal disease (calculated GFR <50% reduced from normal), liver disease (AST or AST > 3 times upper limit of normal), greater than 10 mg of prednisone or equivalent, hypercalcemia, history of easily burned skin after sunlight exposure, taking medications with may cause photosensitivity, history of skin cancer or multiple moles or family history of skin cancer, moderate to severe vitamin D deficiency (25(OH)D ≤ 15 ng/ml).

Physicians at the Emory CF center will be informed about the study. The primary CF doctor of the subject will refer the individual to one of the study investigators for potential recruitment. The principal investigator or co-investigator will meet with the prospective subject to discuss the details of the study. If the subject agrees to participate, they will sign an informed consent form. The subject will provide a blood specimen at the screening visit to determine eligibility for the study including 25-hydroxyvitamin D. If the subject's 25(OH)D level is ≤15 ng/ml (moderate vitamin D deficiency), the subject will be excluded from the study. We have decided to exclude those moderately to severely deficient patients for ethical reasons since these subjects may require more aggressive medical management in correction of vitamin D status.

The subject will then be randomized to either ergocalciferol 50,000 IU once a a week for 12 weeks, cholecalciferol 50,000 IU once a week for 12 weeks, or use of a portable tanning device 5 times a week for 12 weeks. The blood sample obtained for screening will be used to determine baseline 25(OH)D, parathyroid hormone (PTH). This assignment can not be blinded for obvious reasons. Subjects assigned to cholecalciferol or ergocalciferol will be instructed on how to take the pill three times a week. The subjects assigned to the portable tanning machine will be given instructions on how to operate the device.

All subjects will complete a baseline three day food diary to determine daily calcium and vitamin D intake levels. Those subjects already taking calcium supplements will be instructed to take no more than 1500 mg of calcium a day. Those subjects already taking multivitamin supplements will be limited to no more than 800 IU of vitamin D daily. Subjects will be allowed to continue with their usual diet; however, they should limit the number of milk servings to no more than 3 servings a day. Subjects will also be instructed not to travel to sunny climates or visit tanning salons during the study. No restrictions will be made in regards to outdoor activities since minimal vitamin D is made during the winter months. Subjects will return to the CF center 12 weeks after the randomization for repeat blood tests for 25(OH)D and PTH. Every two weeks, our research coordinator will call the subject to discuss compliance with the assigned therapy. In particular, those subjects assigned to pills will be reminded to take the pills weekly. Those subjects assigned to UV light will be asked questions regarding presence of skin erythema, photosensitivity, evidence of tanning and any other potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects seen initially at the Emory CF center between the months of September and December
* Age > 16, both males and females, confirmed cystic fibrosis by genetic testing or sweat testing, FEV1 > 40%.

Exclusion Criteria:

* History of lung transplant or awaiting lung transplantation
* Current hospitalization or greater than 6 hospitalizations/year
* History of malignancy, renal disease (calculated GFR < 50% reduced from normal), liver disease (AST or AST > 3 times upper limit of normal), greater than 10 mg of prednisone or equivalent, hypercalcemia
* History of easily burned skin after sunlight exposure, taking medications with may cause photosensitivity
* History of skin cancer or multiple moles or family history of skin cancer
* Moderate to severe vitamin D deficiency (25(OH)D ≤ 15 ng/ml).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, M.D. Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory CF Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Grossmann RE, Zughaier SM, Liu S, Lyles RH, Tangpricha V. Impact of vitamin D supplementation on markers of inflammation in adults with cystic fibrosis hospitalized for a pulmonary exacerbation. Eur J Clin Nutr. 2012 Sep;66(9):1072-4. doi: 10.1038/ejcn.2012.82. Epub 2012 Jul 18. PMID 22805498
- [Result] Grossmann RE, Zughaier SM, Kumari M, Seydafkan S, Lyles RH, Liu S, Sueblinvong V, Schechter MS, Stecenko AA, Ziegler TR, Tangpricha V. Pilot study of vitamin D supplementation in adults with cystic fibrosis pulmonary exacerbation: A randomized, controlled trial. Dermatoendocrinol. 2012 Apr 1;4(2):191-7. doi: 10.4161/derm.20332. PMID 22928076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please see full manuscript
Pre-assignment Details: Please see full manuscript
Groups:
- Vitamin D3: vitamin D3 50,000 IU weekly
- Vitamin D2: vitamin D2 50,000 IU weekly
- Sunlamp: Use of a sunlamp 5 times a week for 12 weeks.
Period: Overall Study
Arm/Group | Vitamin D3 | Vitamin D2 | Sunlamp
Started | 10 | 10 | 10
Completed | 9 | 10 | 9
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Vitamin D2 | Sunlamp | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (12.5) | 27.9 (11.9) | 33.3 (15.7) | 32.1 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 5 | 5 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: 25-hydroxyvitamin D
Description: This is a marker of vitamin D status
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sunlamp: Weekly use of a sunlamp
Arm/Group | Vitamin D3 | Vitamin D2 | Sunlamp
Number analyzed (Participants) | 9 | 10 | 9
ng/mL | 21.2 (10.3) | 24.4 (10.2) | 28.2 (3.2)

2. Secondary Outcome: Parathyroid Hormone, Serum C-telopeptide, Osteocalcin
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Vitamin D3 | Vitamin D2 | Sunlamp
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No